CLINICAL TRIAL: NCT05945446
Title: A Comparative Study of Serum Galectin-3 Levels Between Placenta Accreta Spectrum and Normal Pregnancies
Brief Title: A Serum Galectin-3 Levels in Placenta Accreta Spectrum Pregnancies
Status: Completed | Type: Observational
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Hasan Energin, Assistant professor doctor, Necmettin Erbakan University
Other Study IDs: ecmettinErbakanUniversity
Record Dates: First submitted 2023-07-06; First posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Placenta Accreta, Third Trimester
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal Pregnancies (control group): Healthy pregnancies with similar gestational age and body mass index with study group.
  Interventions: Diagnostic Test: Galectin 3
- Placenta accreta spectrum pregnancies (study group): 34-36 weeks of gestation. Women diagnosed with Placenta Accreta Spectrum (PAS) were invited to join the study, providing they had no known systemic diseases (e.g. chronic hypertension, diabetes, hypothyroidism, chronic renal-liver diseases, etc.), autoimmune disorders, multiple pregnancies, or the presence of fetal structural and chromosomal anomalies. They also did not have cholestasis of pregnancy, preterm delivery, or evidence of chronic and active infection.
  Interventions: Diagnostic Test: Galectin 3

INTERVENTIONS:
Diagnostic Test: Galectin 3 — Women diagnosed with Placenta Accreta Spectrum (PAS) were invited to join the study, providing they had no known systemic diseases (e.g. chronic hypertension, diabetes, hypothyroidism, chronic renal-liver diseases, etc.), autoimmune disorders, multiple pregnancies, or the presence of fetal structural and chromosomal anomalies. They also did not have cholestasis of pregnancy, preterm delivery, or evidence of chronic and active infection.

SUMMARY:
Placenta Accreta Spectrum (PAS) represents a significant cause of maternal morbidity and mortality, causing complications that surpass those posed by most routine obstetric issues. As such, early detection and proper management of PAS can significantly improve pregnancy outcomes. This study provides an in-depth examination of the serum levels of Galectin-3, a β-galactoside-binding protein, in women experiencing Placenta Accreta Spectrum compared to those with normal pregnancies.

DETAILED DESCRIPTION:
Placenta Accreta Spectrum (PAS) represents a significant cause of maternal morbidity and mortality, causing complications that surpass those posed by most routine obstetric issues. As such, early detection and proper management of PAS can significantly improve pregnancy outcomes. This study provides an in-depth examination of the serum levels of Galectin-3, a β-galactoside-binding protein, in women experiencing Placenta Accreta Spectrum compared to those with normal pregnancies.

Galectin-3 has been implicated in various physiological processes such as cell-cell interaction, cell-matrix adhesion, and immune responses. Moreover, recent evidence suggests an increased level of Galectin-3 is also associated with inflammation, fibrosis, and adverse outcomes in several pathological conditions like cardiovascular diseases and cancer. These multiple roles of Galectin-3 underline its potential implications and predictive ability in many pathological conditions including PAS disease progression during pregnancy.

In obstetric context, research on the role and level of Galectin-3 is sparse. This study aims at filling this gap by comparing the serum Galectin-3 levels in PAS and normal pregnancies. It seeks to investigate whether there is a significant difference between the two cohorts, which could highlight the potential use of Galectin-3 as a possible biological marker in predicting or diagnosing placenta accreta spectrum.

ELIGIBILITY:
Inclusion Criteria:

* PAS diagnosis

Exclusion Criteria:Systemic diseases (e.g. chronic hypertension, diabetes, hypothyroidism, chronic renal-liver diseases, etc.), autoimmune disorders, multiple pregnancies, or the presence of fetal structural and chromosomal anomalies. Cholestasis of pregnancy, preterm delivery, or evidence of chronic and active infection.

-

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Study Population: Women diagnosed with Placenta Accreta Spectrum (PAS) were invited to join the study, providing they had no known systemic diseases (e.g. chronic hypertension, diabetes, hypothyroidism, chronic renal-liver diseases, etc.), autoimmune disorders, multiple pregnancies, or the presence of fetal structural and chromosomal anomalies. They also did not have cholestasis of pregnancy, preterm delivery, or evidence of chronic and active infection.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Galectin 3 | 34-36 weeks of gestation
  Serum Galectin 3 levels

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University Meram Medicine Faculty, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data will be shared if asked for proper reason

REFERENCES:
- [Background] Bojic-Trbojevic Z, Jovanovic Krivokuca M, Vilotic A, Kolundzic N, Stefanoska I, Zetterberg F, Nilsson UJ, Leffler H, Vicovac L. Human trophoblast requires galectin-3 for cell migration and invasion. Sci Rep. 2019 Feb 14;9(1):2136. doi: 10.1038/s41598-018-38374-w. PMID 30765738
- [Background] Pankiewicz K, Szczerba E, Fijalkowska A, Szamotulska K, Szewczyk G, Issat T, Maciejewski TM. The association between serum galectin-3 level and its placental production in patients with preeclampsia. J Physiol Pharmacol. 2020 Dec;71(6). doi: 10.26402/jpp.2020.6.08. Epub 2021 Mar 13. PMID 33727431